CLINICAL TRIAL: NCT06688240
Title: A Multi-center, Single-arm, Prospective Non-interventional Study to Investigate the Safety Profiles and Effectiveness of Liposomal Irinotecan (ONIVYDE®) in Combination with 5-fluorouracil (5-FU) and Leucovorin (LV) in Chinese Patients with Metastatic Pancreatic Cancer As Approval Condition (SEOPAC)
Acronym: SEOPAC
Status: Not yet recruiting | Type: Observational
Sponsor: Servier (Tianjin) Pharmaceutical Co. LTD. (Industry)
Collaborators: Les Laboratoires Servier (Unknown)
Responsible Party: Sponsor
Other Study IDs: SAF-95013-001-CHN
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- prescribed for ONIVYDE treatment according to the ONIVYDE China mainland SmPC: this is a prospective, single-arm, multicenter, open-label and non-interventional study

SUMMARY:
The aim of this phase 4 study is to evaluate the safety profile of ONIVYDE in China mainland.

Primary objective

To characterize the safety of ONIVYDE when used under standard clinical practice in China mainland on the following aspects:

1. Quantify the rate of grade ≥3 neutropenia (primary objective)
2. Serious adverse events and serious adverse drug reactions
3. Adverse events and adverse drug reactions Secondary objective To describe effectiveness in patients receiving ONIVYDE in combination with 5-FU and leucovorin for the treatment of metastatic pancreatic cancer under standard clinical care in China mainland.

(1) Overall survival (2) Overall response (3) Progression free survival (4) Quality of life assessment

ELIGIBILITY:
Inclusion Criteria:

* The adult patient (≥18 years of age) has given written informed consent to participate in the study.
* The patient has been prescribed for ONIVYDE treatment according to the ONIVYDE China mainland SmPC.
* Histologically or cytologically confirmed adenocarcinoma of exocrine pancreas.
* Documented metastatic disease.
* Patient deemed not eligible or failed previous treatment with gemcitabine or gemcitabine containing therapy.

Exclusion Criteria:

* Patients who have experienced a severe hypersensitivity reaction to ONIVYDE or Irinotecan HCL.
* Patients with new or progressive dyspnea, cough, and fever, pending diagnostic evaluation or confirmed diagnostic of interstitial lung disease.
* Pregnant or nursing (lactating) women.
* Patients without highly effective methods of contraception during study treatment until 3 months after the last dose of the study drug, Specially,7 months for women of childbearing potential and 4 months for male with partners of childbearing potential after the last dose of the study drug.
* Other additional exclusions may be applied by the investigator according to the contexts, in order to ensure that the study population will be non-interventional but representative of all eligible subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For a margin of error of 10% and to adjust for 20% dropout, a sample size of 120 patients is needed to produce a two-sided 95% CI when the estimate of proportion (Grade 3 and higher neutropenia) is 55% (Occurrence rate of grade 3 and higher neutropenia is about 55% in Asia patients in NAPOLI-1).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety of ONIVYDE when used under standard clinical practice in China mainland on the following aspects: | From enrolment until 30 days after last ONIVYDE administration
  (1) Quantify the rate of grade ≥3 neutropenia (primary objective)
To characterize the safety of ONIVYDE when used under standard clinical practice in China mainland on the following aspects: | From enrolment until 30 days after last ONIVYDE administration
  (2) Serious adverse events and serious adverse drug reactions
To characterize the safety of ONIVYDE when used under standard clinical practice in China mainland on the following aspects: | From enrolment until 30 days after last ONIVYDE administration
  (3) Adverse events and adverse drug reactions

SECONDARY OUTCOMES:
To describe effectiveness in patients receiving ONIVYDE in combination with 5-FU and leucovorin for the treatment of metastatic pancreatic cancer under standard clinical care in China mainland. | From FPI to 12 months after LPI
  (1) Overall survival
To describe effectiveness in patients receiving ONIVYDE in combination with 5-FU and leucovorin for the treatment of metastatic pancreatic cancer under standard clinical care in China mainland. | From FPI to 12 months after LPI
  (2) Overall response
To describe effectiveness in patients receiving ONIVYDE in combination with 5-FU and leucovorin for the treatment of metastatic pancreatic cancer under standard clinical care in China mainland. | From FPI to 12 months after LPI
  (3) Progression free survival
To describe effectiveness in patients receiving ONIVYDE in combination with 5-FU and leucovorin for the treatment of metastatic pancreatic cancer under standard clinical care in China mainland. | From FPI to 12 months after LPI
  (4) Quality of life assessment(e.g.Karnofsky Performance Status (KPS))

IPD SHARING:
Plan to Share IPD: No